CLINICAL TRIAL: NCT05269628
Title: Mechanisms of Cannabidiol (CBD) in Persons With Multiple Sclerosis (MS): the Role of Sleep and Pain Phenotype
Brief Title: Mechanisms of Cannabidiol in Persons With MS: the Role of Sleep and Pain Phenotype
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tiffany J. Braley, MD, MS (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor-Investigator, Tiffany J. Braley, MD, MS, Associate Professor of Neurology, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HUM00190734; 1R01AT011341-01 (NIH)
Record Dates: First submitted 2022-02-13; First posted 2022-03-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis; Sleep; Pain
Keywords: Cannabidiol
MeSH Terms: conditions — Multiple Sclerosis; Pain | interventions — Cannabidiol; Solutions; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cannabidiol (CBD) (Experimental): Cannabidiol (Epidiolex® 100 mg/mL solution) will initially be prescribed as 50 mg (0.5 mL) twice daily during the first seven days of active treatment (half of full anticipated dose), followed by 100 mg (1 mL) twice daily for the remainder of the treatment interval (full dose).
  PLUS Placebo Tetrahydrocannabinol (TCH) capsules which contain no active ingredients. Matching placebo capsules will be taken twice per day in the same schedule and manner as active dronabinol.
  Interventions: Drug: Cannabidiol (CBD); Drug: Placebo THC
- Tetrahydrocannabinol (THC) (Active Comparator): Tetrahydrocannabinol (Dronabinol capsules) will initially be prescribed as 2.5 mg twice daily during the first seven days of active treatment (half of full anticipated dose), followed by 5 mg twice daily for the following days of active treatment (full dose).
  PLUS Placebo CBD (A matching placebo oral solution to Epidiolex® will be used that consists of all of the excipients in the active solution without the cannabidiol component). The placebo will be dosed in the same schedule and manner as active Epidiolex®.
  Interventions: Drug: Tetrahydrocannabinol (THC); Drug: Placebo CBD
- CBD + THC (Active Comparator): Cannabidiol (Epidiolex® solution) will initially be prescribed as 50 mg (0.5 mL) twice daily during the first seven days of active treatment (half of full anticipated dose), followed by 100 mg (1 mL) twice daily for the remainder of the treatment interval (full dose).
  PLUS Tetrahydrocannabinol (Dronabinol capsules) will initially be prescribed as 2.5 mg twice daily during the first seven days of active treatment (half of full anticipated dose), followed by 5 mg twice daily for the following days of active treatment (full dose).
  Interventions: Drug: Cannabidiol (CBD); Drug: Tetrahydrocannabinol (THC)
- Placebo CBD + Placebo THC (Placebo Comparator): Placebo CBD (A matching placebo oral solution to Epidiolex® will be used that consists of all of the excipients in the active solution without the cannabidiol component). The placebo will be dosed in the same schedule and manner as the active CBD.
  PLUS Placebo Tetrahydrocannabinol (TCH) capsules which contain no active ingredients. Matching placebo capsules will be taken twice per day in the same schedule and manner as active drug.
  Interventions: Drug: Placebo CBD; Drug: Placebo THC

INTERVENTIONS:
Drug: Cannabidiol (CBD) — Epidiolex® dose will be 0.5 mL (50 mg) twice daily during the first seven days of active treatment (half of full anticipated dose), followed by 1 mL (100 mg) twice daily for the remainder of the treatment interval (full dose). If the full dose (100 mg twice daily) is not tolerated by participants, they will have the option of going down to the original half-dose (50 mg twice daily).
  Participants who go back to the half-dose of Cannabidiol (50 mg twice daily) also have the option to request once-per-day dosing with study drug taken at preferred time of day. Participants who request once-per-day dosing will not exceed a total daily dose 100 mg Cannabidiol per day. Participants who are tolerating the full-dose of medication (Cannabidiol 100 mg twice daily) will not be allowed to combine these doses into one daily dose.
  Other Names: Epidiolex® 100 mg/mL solution
  Arms: CBD + THC; Cannabidiol (CBD)
Drug: Tetrahydrocannabinol (THC) — Dronabinol dose will be 2.5 mg twice daily during the first seven days of active treatment (half of full anticipated dose), followed by 5 mg twice daily for the remainder of the treatment interval (full dose). If the full dose (5 mg twice daily) is not tolerated by participants, they will have the option of going down to the original half-dose (2.5 mg twice daily).
  Participants who go back to the half-dose of Dronabinol (2.5 mg twice daily) also have the option to request once-per-day dosing with study drug taken at preferred time of day. Participants who request once-per-day dosing will not exceed a total daily dose 5 mg Dronabinol per day. Participants who are tolerating the full-dose of medication (Dronabinol 5 mg BID) will not be allowed to combine these doses into one daily dose.
  Other Names: Marinol®, dronabinol capsules
  Arms: CBD + THC; Tetrahydrocannabinol (THC)
Drug: Placebo CBD — Placebo solution will be taken twice per day, using the same dosing regimen as described for Epidiolex®.
  Arms: Placebo CBD + Placebo THC; Tetrahydrocannabinol (THC)
Drug: Placebo THC — Placebo capsules will be taken twice per day in the same schedule and manner as active dronabinol.
  Arms: Cannabidiol (CBD); Placebo CBD + Placebo THC

SUMMARY:
The purpose of this research study is to compare the effects of cannabidiol (CBD), tetrahydrocannabinol (THC), or both, on sleep and pain in persons with multiple sclerosis (MS). Little is known about how CBD and/or THC may help sleep, reduce pain, or perhaps even treat pain through better sleep.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clinically definite MS (those who are on a disease modifying therapy must be on a stable dose without evidence of liver toxicity for at least 3 months);
2. Presence of chronic pain defined as moderate to severe pain for at least 3 months, based on a 0-10 numeric rating scale (NRS);
3. Willingness to maintain stable analgesic regimen during study period;
4. Recent serum aspartate transaminase, alanine transaminase, and bilirubin testing within 90 days of screening;

Exclusion Criteria:

1. Current shift work sleep disorder, or narcolepsy diagnosed with polysomnography and multiple sleep latency test;
2. History of MS relapse within the last 30 days prior to screening (participants will be considered eligible after the 30-day window);
3. Pain due to cancer;
4. Pregnancy or breastfeeding;
5. Current cannabinoid use (participants may be reconsidered for inclusion after 30-day washout) and/or unwillingness to abstain from cannabinoids in any form from 30 days prior to the study of the study drugs and until the last follow up phone call at the end of the study (30 - 37 days after taking the last dose of the study drug).
6. Unwillingness to use contraception from screening until the end of drug treatment
7. Current suicidal ideation (SI) with intent and/or plan; these individuals will be assessed by a study psychologist and referred for urgent mental health treatment as indicated;
8. Current severe depression as indicated by a PHQ-9 score of ≥ 17 that includes indicators of significant depressed mood (sum of items #1 and #2 ≥ 5).
9. History of mania or schizophrenia diagnosis
10. Known hypersensitivity to cannabinoids in general, or Epidiolex® or Dronabinol specifically or its excipients (e.g., sesame oil)
11. History of the following cardiovascular conditions: recent myocardial infarction or stroke (last 6 months prior to screening), unstable angina, left ventricular hypertrophy, mitral valve prolapses, severe coronary artery disease, NYHA class III or IV congestive heart failure.
12. History severe hepatic impairment (must have blood AST ≤ 2.0x ULN, ALT ≤ 2,0x ULN, and bilirubin ≤ 1.5x ULN within the last 90 days (AST, ALT, bilirubin testing will be required within 90 days of screening);
13. History of seizure disorder (recurrent, unprovoked seizures not explained by a known reversible cause) or history of certain types of head injury that could cause an increased risk of seizures;
14. History of prescription or illicit drug abuse (such as cocaine, amphetamine, methamphetamine, heroin);
15. Current risk for alcohol misuse as indicated by a score of ≥ 8 on the Alcohol Use Disorders Identification Test (AUDIT) self-report measure.
16. Current warfarin, valproate or clobazam use.
17. Current use of known moderate or strong inhibitors of CYP3A4 [topical ketoconazole, and temporary (<= 4 week) oral courses of clarithromycin, fluconazole and itraconazole will be allowed].
18. Current use of strong inducers of CYP3A4 or CYP2C19 (does not include glucocorticoids or modafinil/armodafinil, which are permitted),
19. Current use of moderate or strong inhibitors/inducers of CYP2C9, and narrow therapeutic index drugs (e.g., cyclosporine, amphotericin B).
20. Current use of known non-minor Sensitive CYP2C19 Substrates, with the exception of some proton pump inhibitors (e.g., esoprazole, omeprazole)), periodic self-limited courses of diazepam (e.g., for MRI sedation) and submaximal doses of some antidepressant class medications (e.g., citalopram, and escitalopram), which will be permitted by the discretion of the treating neurologist PI.
21. Refusal to avoid grapefruit or grapefruit products during the study treatment interval.
22. Current use of opioids (tramadol permitted).
23. Employed as a commercial driver or employed in an occupation that involves extreme heights or use of heavy machinery.
24. History of car crashes or near-crashes due to untreated sleepiness that has led to near-misses in the past 6 months.
25. Cognitive dysfunction as indicated by >=3 errors on the six-item cognitive screener
26. Expanded Disability Status Scale (EDSS) score >=8.0.
27. Blood pressure at screening above 180 mmHg systolic and/or 120 mmHg diastolic, or below 90 mmHg systolic and or 60 mmHg diastolic, or history of syncope related to orthostatic hypotension;
28. Resting heart rate at screening less than 50 bpm or greater than 100 bpm;
29. Any other treatment or medical, neurological, sleep, or psychiatric condition that, in the opinion of the investigators, could affect participant safety or eligibility.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in sleep bout length | Baseline, 12 weeks
  Measured with in-laboratory polysomnography, reported as average length of continuous bouts of sleep, for each sleep stage and total sleep (in minutes).
Change in Walsh Spectral Entropy | Baseline, 12 weeks
  Measured with in-laboratory polysomnography, computed from EEG sleep stage data to quantify hypnogram regularity (dimensionless, values range from 0-1)
Change in Transition Entropy | Baseline, 12 weeks
  Measured with in-laboratory polysomnography. Entropy measure computed from sleep stage transition matrix that quantifies hypnogram regularity (dimensionless, values range from 0-1)
Change of center of activity | Baseline, 12 weeks
  Measured with in-laboratory polysomnography. Weighted mean temporal location over the night of all 30 second epochs scored as N3 and Rapid eye movement (REM) sleep
Change in sleep rhythmicity | Baseline, 12 weeks
  Measured by actigraphy. Probability of being in the same sleep/wake state 24h apart
Change in sleep regularity | Baseline, 12 weeks
  Measured by actigraphy in hours.
Change in sleep continuity and duration | Baseline, 12 weeks
  Measured by actigraphy in minutes to obtain time in wakefulness after sleep onset (WASO) and total sleep time.

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Braley, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No